CLINICAL TRIAL: NCT05846373
Title: Effect of Nicotinic Acid as add-on Therapy in Patients Receiving β Blocker for Prophylaxis of Moderate to Severe Migraine: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Nicotinic Acid as Add on Therapy in Patients Receiving β Blocker for Prophylaxis of Moderate to Severe Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Hudia Ta-din, MBBS, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSMMU/2022/11548
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-01

CONDITIONS: Migraine Prophylaxis
MeSH Terms: interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotinic Acid Extended-release tablet 500 mg arm (Active Comparator): This arm includes 22 Migraine patients receiving beta blocker
  Interventions: Drug: Nicotinic Acid 500 MG Extended Release Oral Tablet
- Nicotinic Acid Extended-release tablet 1000 mg arm (Active Comparator): This arm includes 22 Migraine patients receiving beta blocker
  Interventions: Drug: Nicotinic Acid 1000 MG Extended Release Oral Tablet
- Control arm (Placebo Comparator): This arm includes 22 Migraine patients receiving beta blocker
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotinic Acid 500 MG Extended Release Oral Tablet — Nicotinic acid 500 mg for 12 weeks
  Other Names: Niacin
  Arms: Nicotinic Acid Extended-release tablet 500 mg arm
Drug: Nicotinic Acid 1000 MG Extended Release Oral Tablet — Nicotinic acid 1000 mg per day for 11 weeks, titrated from 500 mg/day for 1 week
  Other Names: Niacin
  Arms: Nicotinic Acid Extended-release tablet 1000 mg arm
Other: Placebo — Placebo 1000 mg per day for 11 weeks, titrated from 500 mg/day for 1 week
  Arms: Control arm

SUMMARY:
This is a prospective single center, randomized, double-blind, 3 arm placebo-controlled study in subjects with migraine headache requiring prophylactic treatment. The patients will be randomized to receive Nicotinic Acid Extended-release tablet 500 mg or 1000 mg or placebo for 12 weeks. The safety and efficacy outcome measures will be assessed at baseline and 12 weeks.

DETAILED DESCRIPTION:
Migraine is "a common episodic neurological disorder with complex pathophysiology that manifests as recurrent attacks of typically throbbing and unilateral, often severe headache with certain associated features such as nausea, phonophobia, and photophobia". Worldwide, estimated prevalence was 13.8% to 15%. Quality of life of a migraine patient is extremely low and migraine badly hampers one's physical, emotional, and social efficiency and disrupt familial, social and professional relationships. Diagnosis is solely clinical depending on characteristics of headache and associated symptoms. Neuroimaging can be done only when exclusion of another cause of headache is needed.

Exact etiology and pathophysiology of migraine is unknown and multifactorial. There are several hypotheses of migraine pain generation. Local dilatation of intracranial and extracerebral vessels activate trigeminal nerve surrounding cerebral and meningeal vasculature. Migraine pain starts from the activation of trigeminovascular system. Afferent fibers innervating cerebral and meningeal vessels project to central nervous system and releases vasoactive peptides and inflammatory mediators. Some important mediators like Calcitonin gene related peptide (CGRP), NO, Substance P play role in inflammation and vasodilatation. Then sensitization and discharge of thalamic neuron and subsequent projection to sensory cortical neurons occurs. Thus, pain perception is received in migraine.

In studies, elevated levels of C reactive protein (CRP) and Transforming growth factor β (TGF-β) provides evidence of neuroinflammation. In migraine, impairment of cerebral mitochondrial energy metabolism and oxidative stress occurs. As a result, abnormalities in cerebral vasculature results in Cortical Spreading Depression (CSD).

Niacin, which is known as nicotinic acid or Vitamin B3 is the precursor of Nicotinamide Adenine Dinucleotide (NAD) or Nicotinamide Adenine Dinucleotide Phosphate (NADP). From dietary tryptophan, through kynurenine pathway, NAD is produced, and rest 1% tryptophan is catabolized to form serotonin (5- hydroxytryptamine/ 5-HT). Migraine is a serotonin deficient condition. It has been estimated that, dietary intake of Niacin is low in migraine patients.

Niacin supplementation provides enough NAD to inhibit Kynurenine pathway and accelerate production of 5-HT from tryptophan. Serotonin acting on 5-HT1 receptor, causes vasoconstriction. It may activate nerve endings in cerebral microcirculation and sensitize them to vasodilatory kinins. Serotonin also inhibits synthesis, release of NO, glutamate, Calcitonin gene-related peptide (CGRP). As a result, inhibition of afferent pain transmission and prevention of neuroinflammation occurs. Niacin also reduces inflammation evidenced by decrease level of pro inflammatory cytokines like IL-6, IL-1β, TNF α, high-sensitivity C-reactive protein (hs-CRP). Increasing level of Niacin also improves brain energy deficiency, and has potent antioxidant properties, which may be helpful in migraine prevention. However, more prospective investigations are necessary to validate niacin's preventive effect on migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from migraine with or without aura according to International ICHD 3 criteria
2. Patients with 4-15 qualified migraine attacks per month during the four weeks of the Baseline Phase
3. History of headache for at least 1 year
4. Age at onset of migraine should be less than 50 years
5. Headache intensity: Moderate to severe (Visual analogue scale score at least 3)
6. Consuming one β Blocker as prophylaxis

Exclusion Criteria:

1. Pregnancy and lactation
2. Known case of any hepatic, psychiatric diseases except depression, diabetes mellitus (DM), gout, peptic ulcer disease
3. Known hypersensitivity to niacin
4. Consumption of certain drugs Lipid lowering agents Antiplatelet and Anticoagulants Antihypertensive medications Alcohol or other abusive drugs
5. Plasma Nicotinic acid level > 8.45 µg/mL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Migraine days/4 weeks | Baseline to week 12
  Mean change from baseline in migraine days/4 weeks from baseline to weeks 9-12

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score | Baseline to week 12
  Changes of mean VAS Score from baseline to weeks 9 - 12. The average migraine attack severity will be calculated using the sum of the severity of migraine attacks, divided by the number of qualified migraine attacks. The scale of severity for each migraine attack ranges from 0 to 10, with higher scores indicating increased migraine severity.
Migraine Specific Quality of Life questionnaire version 2.1 (MSQ V. 2.1) | Baseline to week 12
  Changes of mean MSQ V. 2.1 score from baseline to weeks 9 -12. The MSQ V. 2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains; Role function restrictive (RR), Role function preventive (RP), Emotional function (EF) consist of 7, 4 and 3 items respectively. Score ranges from 0 - 100 in each domain. The higher scores indicate better outcome.
Frequency of use of acute migraine specific medications in the last 4 weeks | Baseline to week 12
  Changes in number of days receiving migraine aborting medication/(s) from baseline to weeks 9-12
hs-CRP | Baseline to week 12
  Change in hs-CRP level from baseline to week 12

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh